CLINICAL TRIAL: NCT06708403
Title: Effects of Judo- Specific Injury Prevention Exercise Programme on Performance in Recreational Judo Athletes
Brief Title: Effects of Judo- Specific Injury Prevention Exercise Programme Judo Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/RCR & AHS/24/0418
Record Dates: First submitted 2024-11-18; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: Judo; Sports injury; Martial art; Agility; Plyometric exercise; Strength; IPPON
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Judo-Specific Injury Prevention Exercise Program (Experimental): 18 participants will be in the experimental group, following a judo-specific injury prevention exercise protocol for six weeks (three sessions per week).
  Baseline and post-intervention measurements will evaluate judo-specific skills, agility, balance, and overall performance.
  The intervention will include:
  Warm-up exercises tailored for injury prevention Strength and conditioning exercises specific to judo movements Drills focusing on balance, agility, and coordination Gradually progressive intensity over six weeks
  Interventions: Other: Judo-Specific Injury Prevention Exercise Program
- Regular Judo Training (No Intervention): 18 participants will be in the control group, continuing their regular judo training sessions without any additional intervention.
  The same performance metrics will be measured at baseline and post-intervention.
  The control group will continue their regular training sessions as guided by their judo coaches, with no alterations.

INTERVENTIONS:
Other: Judo-Specific Injury Prevention Exercise Program — The intervention includes a structured program designed specifically for judo athletes to prevent injuries and enhance performance. The program consists of warm-up exercises, strength and conditioning drills, balance improvement exercises, agility training, and sport-specific movements. It is delivered over six weeks, with participants completing three sessions per week. Each session is progressively tailored to improve overall motor skills, prevent overuse injuries, and enhance judo-specific abilities.
  Arms: Judo-Specific Injury Prevention Exercise Program

SUMMARY:
The study aimed to determine whether the judo-specific injury prevention exercise program had a significant positive effect on the performance of recreational judo athletes, with a particular focus on those employing the ippon technique.

DETAILED DESCRIPTION:
The significant results obtained from our study are considered to be originated from the duration, scope, frequency, severity and content of training.

ELIGIBILITY:
Inclusion Criteria:

* Recreational judo athletes aged 18 to 35 years.
* Participants with at least one year of regular participation in recreational judo Athletes with no existing major musculoskeletal injuries or chronic health conditions that would limit their ability to participate in the prescribed exercise program.
* Participants willing to provide informed consent and commit to the duration of the study, including regular attendance at training sessions and data collection activities.
* Athletes engaging in judo training at least twice a week.

Exclusion Criteria:

* Athletes below 18 or above 35 years of age.
* Novice judo practitioners with less than one year of regular training.
* Individuals with a history of significant musculoskeletal injuries in the past six months or chronic conditions affecting their ability to participate fully.
* Participants unwilling or unable to provide informed consent or commit to the study requirements.
* Athletes participating in judo training less than twice a week, as they may not represent a group with sufficient exposure to the injury prevention program.
* Professional or highly competitive judo athletes, as their training regimens and performance levels may differ significantly from recreational athletes.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Injury Incidence and Severity | Weekly assessments during the 6-week intervention
  The OSTRC Overuse Injury Questionnaire will be used to measure the incidence and severity of overuse injuries in participants. This tool evaluates pain, function, and participation limitations experienced during training and judo activities.
  Parameters Assessed:
  Presence of pain (location and intensity) Impact on training participation Functional limitations caused by pain or injury
Judo-Specific Performance Assessment | Baseline (pre-intervention) and 6 weeks (post-intervention)
  Performance in judo-specific skills will be assessed through a task-specific checklist, evaluating speed, accuracy, and execution of techniques during a simulated judo match.
Agility Test Score | Baseline (pre-intervention) and 6 weeks (post-intervention).
  The change in agility will be assessed using the Illinois Agility Test. The test will measure the time (in seconds) taken to complete the agility course.
Balance Assessment | Baseline (pre-intervention) and 6 weeks (post-intervention)
  The improvement in balance will be assessed using the Balance Error Scoring System (BESS), measuring the number of errors in static and dynamic postures.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- The University Of Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franchini E, Julio UF, Panissa VL, Lira FS, Gerosa-Neto J, Branco BH. High-Intensity Intermittent Training Positively Affects Aerobic and Anaerobic Performance in Judo Athletes Independently of Exercise Mode. Front Physiol. 2016 Jun 28;7:268. doi: 10.3389/fphys.2016.00268. eCollection 2016. PMID 27445856
- [Background] Kang H. Sample size determination and power analysis using the G*Power software. J Educ Eval Health Prof. 2021;18:17. doi: 10.3352/jeehp.2021.18.17. Epub 2021 Jul 30. PMID 34325496
- [Background] Honorato RC, Franchini E, Lara JPR, Fonteles AI, Pinto JCBL, Mortatti AL. Differences in Handgrip Strength-Endurance and Muscle Activation Between Young Male Judo Athletes and Untrained Individuals. Res Q Exerc Sport. 2021 Mar;92(1):1-10. doi: 10.1080/02701367.2019.1699233. Epub 2020 Feb 5. PMID 32023202
- [Background] Kowalczyk M, Zgorzalewicz-Stachowiak M, Blach W, Kostrzewa M. Principles of Judo Training as an Organised Form of Physical Activity for Children. Int J Environ Res Public Health. 2022 Feb 9;19(4):1929. doi: 10.3390/ijerph19041929. PMID 35206114
- [Background] Kons RL, Orssatto LBDR, Sakugawa RL, da Silva Junior JN, Diefenthaeler F, Detanico D. Effects of stretch-shortening cycle fatigue protocol on lower limb asymmetry and muscle soreness in judo athletes. Sports Biomech. 2023 Sep;22(9):1079-1094. doi: 10.1080/14763141.2020.1779335. Epub 2020 Jul 9. PMID 32644009
- [Background] Tsai CL, Chien CY, Pan CY, Tseng YT, Wang TC, Lin TK. Effects of long-term Tai Chi vs. aerobic exercise on antioxidant activity and cognitive function in individuals with Parkinson's disease. Behav Brain Res. 2025 Jan 5;476:115274. doi: 10.1016/j.bbr.2024.115274. Epub 2024 Sep 25. PMID 39332640
- [Background] Garbeloto F, Miarka B, Guimaraes E, Gomes FRF, Tagusari FI, Tani G. A New Developmental Approach for Judo Focusing on Health, Physical, Motor, and Educational Attributes. Int J Environ Res Public Health. 2023 Jan 27;20(3):2260. doi: 10.3390/ijerph20032260. PMID 36767628
- [Background] Lee TI, Wang MY, Huang BR, Hsu CY, Chien CY. Effects of Psychological Capital and Sport Anxiety on Sport Performance in Collegiate Judo Athletes. Am J Health Behav. 2022 Apr 20;46(2):197-208. doi: 10.5993/AJHB.46.2.9. PMID 35501965
- [Background] Detanico D, Kons RL, Fukuda DH, Teixeira AS. Physical Performance in Young Judo Athletes: Influence of Somatic Maturation, Growth, and Training Experience. Res Q Exerc Sport. 2020 Sep;91(3):425-432. doi: 10.1080/02701367.2019.1679334. Epub 2020 Jan 6. PMID 31906807
- [Background] Kajmovic H, Karpljuk D, Kapo S, Simenko J. Comparison of Individual Penalties According to Gender and Weight Categories of Elite Judo Athletes from Four World Championships. Biology (Basel). 2022 Aug 29;11(9):1284. doi: 10.3390/biology11091284. PMID 36138762
- [Background] Ouergui I, Franchini E, Selmi O, Levitt DE, Chtourou H, Bouhlel E, Ardigo LP. Relationship between Perceived Training Load, Well-Being Indices, Recovery State and Physical Enjoyment during Judo-Specific Training. Int J Environ Res Public Health. 2020 Oct 11;17(20):7400. doi: 10.3390/ijerph17207400. PMID 33050671
- [Background] Kons RL, Athayde MSDS, Antunes L, Lopes JSS, Detanico D. Injuries in Judo Athletes With Disabilities: Prevalence, Magnitude, and Sport-Related Mechanisms. J Sport Rehabil. 2022 May 4;31(7):904-910. doi: 10.1123/jsr.2021-0352. Print 2022 Sep 1. PMID 35508305
- [Background] von Gerhardt AL, Vriend I, Verhagen E, Tol JL, Kerkhoffs GMMJ, Reurink G. Systematic development of an injury prevention programme for judo athletes: the IPPON intervention. BMJ Open Sport Exerc Med. 2020 Sep 29;6(1):e000791. doi: 10.1136/bmjsem-2020-000791. eCollection 2020. PMID 33033621
- [Background] von Gerhardt AL, Reurink G, Kerkhoffs GMMJ, Verhagen E, Krabben K, Mooren J, Gal JSI, Brons A, Joorse R, van den Broek B, Kemler E, Tol JL. Effectiveness of a judo-specific injury prevention programme: a randomised controlled trial in recreational judo athletes. Br J Sports Med. 2023 Apr;57(8):450-456. doi: 10.1136/bjsports-2022-105869. Epub 2023 Jan 30. PMID 36717214